CLINICAL TRIAL: NCT06428357
Title: Efficacy of Recombinant Bovine Lactoferrin (rbLf) in Iron Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: TurtleTree Labs Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 23-3039
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Exercise Performance
Keywords: Iron regulation
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Females: Recombinant Bovine Lactoferrin (rbLf), then Bovine milk derived Lactoferrin (Experimental): After a 2-week run-in period, this arm will begin treatment with recombinant bovine lactoferrin for 4 weeks and following a 2-week washout start bovine milk derived lactoferrin for 4 weeks.
  Interventions: Dietary Supplement: Recombinant Bovine Lactoferrin; Dietary Supplement: Bovine Milk-Derived Lactoferrin
- Females: Bovine milk derived lactoferrin (cmdLf), then Recombinant bovine lactoferrin (Active Comparator): After a 2-week run-in period, this arm will begin treatment with bovine milk derived lactoferrin and then following a 2-week washout start recombinant bovine lactoferrin for 4 weeks.
  Interventions: Dietary Supplement: Recombinant Bovine Lactoferrin; Dietary Supplement: Bovine Milk-Derived Lactoferrin
- Males: Recombinant Bovine Lactoferrin (rbLf), then placebo (Active Comparator): After a 2-week run-in period, this arm will begin treatment with recombinant bovine lactoferrin for 4 weeks and following a 2-week washout start placebo for 4 weeks.
  Interventions: Dietary Supplement: Recombinant Bovine Lactoferrin; Dietary Supplement: Placebo
- Males: Placebo, then recombinant bovine lactoferrin (rbLf) (Placebo Comparator): After a 2-week run-in period, this arm will begin treatment with placebo for 4 weeks and following a 2-week washout start recombinant bovine lactoferrin for 4 weeks.
  Interventions: Dietary Supplement: Recombinant Bovine Lactoferrin; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Recombinant Bovine Lactoferrin — Participants will take a single dose equal to 3 capsules daily before a meal for 4 weeks. Meal timing is not controlled.
Dietary Supplement: Bovine Milk-Derived Lactoferrin — Participants will take a single dose equal to 3 capsules daily before a meal for 4 weeks. Meal timing is not controlled.
  Arms: Females: Bovine milk derived lactoferrin (cmdLf), then Recombinant bovine lactoferrin; Females: Recombinant Bovine Lactoferrin (rbLf), then Bovine milk derived Lactoferrin
Dietary Supplement: Placebo — Participants will take a single dose equal to 3 capsules daily before a meal for 4 weeks. Meal timing is not controlled.
  Other Names: Sugar Pill
  Arms: Males: Placebo, then recombinant bovine lactoferrin (rbLf); Males: Recombinant Bovine Lactoferrin (rbLf), then placebo

SUMMARY:
Overall Objective: To determine the efficacy of rbLf supplementation in a healthy adult population, specifically with regard to iron regulation (primary), gut health (secondary), and immune function (secondary). Purpose: The purpose of this study is to determine the effects of rbLf on iron regulation, exercise performance, gut health, and immune function as compared to cow's milk derived bLf.

Participants: To account for an approximate ~10% dropout rate (and rounding up to ensure equal number of enrolled participants per group), n=25 per group for males (N=50) and n=30 per group for females (N=60) will be enrolled for a total sample size of N=110.

Procedures: Participation in this study will include 6 in-person visits over 14 weeks. Anemia will be checked and excluded at the first visit using a single finger prick, followed by a 10-20 min exercise test on a treadmill to evaluate exercise capacity. On visit 2 participants will perform three 3-15 minute exercise tests on a treadmill with rest in between each test in order to determine exercise performance. A finger prick will be performed before and after each run to determine lactate levels. After visits 2 participants will be randomized to their respective supplement group recombinant Bovine Lactoferrin supplement (rbLf) (Male and Fame), a bovine-milk derived Lactoferrin supplement (Female), or a placebo (Male) once daily for 4 weeks. Blood samples will be obtained prior to and after each supplement phase to determine change in iron levels and red blood cell capacity. After a 2-week washout participants will return to complete the same testing outcomes and will receive the subsequent supplement. At visit 6 a final blood sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18-42 years
* Body mass index less than 35 kg/m^2
* Finger prick hemoglobin levels fitting within "normal range"

  * Males: 14-18g/dL
  * Females: 12-16g/dL
* Active: meeting American College of Sports Medicine exercise guidelines or exercising more than 2 days per week of

  ● For females specifically:
* Pre-menopausal: experiencing a regular period with no signs of perimenopause or menopause.

Exclusion Criteria:

* Clinically diagnosed iron-deficiency anemia, pagophagia, hemochromatosis, or other blood or iron related medical conditions.
* Allergy or intolerance to milk, egg, soy, peanut, wheat, coconut, or almond dairy
* Smokers or vapers of nicotine or nicotine products
* Immunocompromised or diagnosed with Type I or II diabetes
* Irritable Bowel Disease, Crohn's disease, Celiacs
* Bowel movements less than three times per week, or clinically constipated
* Oral contraceptive users that have combined iron supplementation, or non-monophasic oral contraceptive users.
* Pregnant or nursing
* Chronic eczema or clinically diagnosed asthma.
* Current antibiotic use or antibiotic use within the past 6 weeks
* If flu, corona virus, or cold occurs, subject will remain in the study with their original scheduled visits, but immune values will be excluded.
* Vegan (due to supplement ingredients).

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Change in serum iron (mcg/dL) | baseline to 4 weeks
  change in serum blood values obtained before and after supplementation
Change in ferritin iron (ng/mL) | baseline to 4 weeks
  change in blood values obtained before and after supplementation
Change in red blood cell count (trillion cells/L) | baseline to 4 weeks
  change in blood values obtained before and after supplementation
change in iron binding capacity (mcg/dL) | baseline to 4 weeks
  change in blood values obtained before and after supplementation

SECONDARY OUTCOMES:
change in time to exhaustion running (seconds) | baseline to 4 weeks
  change in treadmill running to exhaustion before and after supplementation
change on tumor necrosis factor-a (pg/mL) | baseline to 4 weeks
  change in blood values obtained before and after supplementation
change in interleukin-6 (pg/ml) | baseline to 4 weeks
  change in blood values obtained before and after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina. Additionally, clear aims and scope of the data request must be included.
Supporting Information: Study Protocol
Time Frame: 9-24 Months after publication
Access Criteria: Clear specific study aims and ethics approval must be present.